CLINICAL TRIAL: NCT01090245
Title: Using Incentives to Improve Parolee Participation and Attendance in Community Tx
Brief Title: Using Incentives to Improve Parolee Participation and Attendance in Community Treatment
Acronym: PIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Michael Prendergast, Research Historian, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R01DA025627-01A1 (NIH)
Record Dates: First submitted 2010-03-16; First posted 2010-03-19 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Substance Abuse; HIV Infections
Keywords: contingency management; substance abuse treatment; criminal justice populations; substance abuse treatment retention; HIV prevention in criminal justice settings; voucher based reinforcement therapy; Parole treatment admission for substance abusing parolees; Parole treatment retention for substance abusing parolees; HIV testing and counseling for substance abusing parolees
MeSH Terms: conditions — Substance-Related Disorders; HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Attendance Information Group (Active Comparator): Participants in the Attendance Information Group will receive an individual information session along with a pamphlet describing the benefits of remaining in treatment after release from prison and on the benefits of HIV prevention and testing. In addition, they will receive the standard treatment offered by the Walden House Los Angeles program.
  Interventions: Behavioral: Information
- Attendance Incentive Group (Experimental): Participants in the Attendance Incentive Group could receive up to $841.50 in incentives for their treatment attendance and the standard treatment offered by the Walden House Los Angeles program.
  Interventions: Behavioral: Contingency management: voucher/monetary incentives for treatment attendance

INTERVENTIONS:
Behavioral: Contingency management: voucher/monetary incentives for treatment attendance — Contingency management: Escalation with reset for non-attendance. Daily. Up to $841.50 in incentives for treatment attendance.
  Arms: Attendance Incentive Group
Behavioral: Information — Attendance Information Group will receive an individual information session along with a pamphlet describing the benefits of remaining in treatment after release from prison and on the benefits of HIV prevention and testing.
  Arms: Attendance Information Group

SUMMARY:
Under funding from the National Institute on Drug Abuse, the UCLA Integrated Substance Abuse Programs (ISAP), in collaboration with Walden House and the California Department of Corrections and Rehabilitation, is conducting a five-year study that will involve a randomized test of the use of incentives with parolees in a community-based residential substance abuse treatment program to increase treatment admission and treatment retention, and thereby increase the likelihood of improved outcomes. Study participants will be recruited from clients in a prison-based treatment program who have a referral to the Walden House community program. The Admission Phase of the study assesses the effect of an incentive (voucher) on enrolling in the Walden House program. The Attendance Phase assesses the effect of incentives on treatment attendance and on post-treatment drug use, crime, and psychosocial behaviors, including HIV risk behaviors. In addition, an incentive protocol will test whether an incentive will encourage participation in HIV testing and counseling. The intervention will last for six months.

Hypothesis 1. The use of incentives will significantly increase subject enrollment in community treatment.

Hypothesis 2. The use of incentives will significantly increase subject retention in community treatment.

Huypothesis 3. The use of incentives will significantly increase subject participation in HIV testing and counseling.

Study participants will be interviewed at baseline and at 12 months following the intervention. Treatment and criminal justice data will be obtained. Data on acceptability, satisfaction, and sustainability will be collected from focus groups with staff and clients.

DETAILED DESCRIPTION:
A considerable body of research indicates that prison-based treatment followed by continuing treatment in the community is effective in reducing drug abuse and crime among drug-abusing offenders. However, the impact of providing treatment is less than optimal because offenders often fail to follow through on treatment referrals, leave treatment early, or have poor engagement in treatment activities. In particular, participation in prison-based treatment alone is seldom effective in reducing drug use or recidivism unless it is followed by participation in community treatment. For correctional systems that provide a continuum of care model from prison to community, low rates of admission and retention result in poor outcomes and poor resource utilization. One way to address this problem is to provide incentives to parolees for community treatment participation. Although research supports the effectiveness of behavioral reinforcement, mainly in the form of contingency management (CM), for general substance abuse populations, CM has not yet been tested or adapted for use in community-based programs for offender populations, particularly to encourage treatment attendance.

In addition, recent research has documented elevated rates of HIV infection among incarcerated populations compared to the general population, with prevalence of HIV among inmates in US prisons being estimated to be 6 to 10 times higher than in the general population. Upon release from prison, parolees often immediately resume high-risk behaviors that they engaged in prior to incarceration. Because of the high level of exposure to HIV infection that accompanies drug use, particularly by injection, drug treatment programs for high-risk offenders can serve as a valuable setting for preventing the spread of HIV, both through HIV prevention/education activities and through access to HIV testing and counseling.

Under funding from the National Institute on Drug Abuse, the UCLA Integrated Substance Abuse Programs (ISAP), in collaboration with Walden House and the California Department of Corrections and Rehabilitation, is conducting a five-year study that will involve a randomized test of the use of incentives with parolees in a community-based residential substance abuse treatment to increase treatment admission and treatment retention, and thereby increase the likelihood of improved outcomes. Study participants will be recruited from clients in a prison-based treatment program who have a referral to the Walden House community program. The Admission Phase of the study assesses the effect of an incentive (voucher) on enrolling in the Walden House program. The Attendance Phase assesses the effect of incentives on treatment attendance and on post-treatment drug use, crime, and psychosocial behaviors, including HIV risk behaviors. In addition, an incentive protocol will test whether an incentive will encourage participation in HIV testing and counseling. The intervention will last for six months.

Hypothesis 1. The use of incentives will significantly increase subject enrollment in community treatment.

Hypothesis 2. The use of incentives will significantly increase subject retention in community treatment.

Huypothesis 3. The use of incentives will significantly increase subject participation in HIV testing and counseling.

Study participants will be interviewed at baseline and at 12 months following the intervention. Treatment and criminal justice data will be obtained. Data on acceptability, satisfaction, and sustainability will be collected from focus groups with staff and clients.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* English speaking
* Within one month of parole
* Able to provide informed consent to participate in the study
* Received a referral to the Walden House Los Angeles Transitional Treatment Center

Exclusion Criteria:

* Potential subjects will be excluded from participating if they have serious cognitive problems that preclude their ability to provide informed consent or understanding of the questionnaire items, if they are a sexually violent predator or a child molester or if they have severe mental health problems.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2010-04; Primary Completion 2014-01 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Community treatment admission | Within 7 days of release to parole
Community treatment retention | 6 months
Participation in HIV testing and counseling | 2 months

SECONDARY OUTCOMES:
Substance abuse | 18 months after release from prison
Arrest and reincarceration | 18 months after release from prison
psychosocial: employment, education, family relationships, psychological functioning, and HIV risk | 18 months after release from prison
  employment, education, family relationships, psychological functioning, and HIV risk

CONTACTS AND LOCATIONS:
Overall Officials: Michael L Prendergast, Ph.D., Principal Investigator — University of California, Los Angeles; Elizabeth A Hall, Ph.D., Study Director — University of California, Los Angeles

REFERENCES:
- [Result] Saxena P, Hall EA, Prendergast M. A Randomized Study of Incentivizing HIV Testing for Parolees in Community Aftercare. AIDS Educ Prev. 2016 Apr;28(2):117-27. doi: 10.1521/aeap.2016.28.2.117. PMID 27459163